CLINICAL TRIAL: NCT03450785
Title: Study About the Incidence and Risk Factors of the Central Line Catheter Related Right Internal Jugular Vein Thrombosis in Pediatric Patients
Brief Title: Incidence and Risk Factors of Central Line Catheter Related Thrombosis
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Other Study IDs: 1801-152-922
Record Dates: First submitted 2018-02-22; First posted 2018-03-01 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Central Line Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ultrasound examination — Doppler ultrasound examinations from the thyroid cartilage level to the supraclavicular region were used after CVC placement and on each of the following days until the catheter was removed.

SUMMARY:
Central venous catheters are frequently used for monitoring haemodynamic status and rapidly delivering fluid therapy during the peri- and postoperative periods. Indwelling central venous catheters are typically used 7-14 days postoperatively for additional monitoring and treatment, but patients may develop asymptomatic catheter-related thrombosis, leading to life-threatening pulmonary embolism and death. Early detection helps to avoid such complications. This prospective observational study investigated the risk factors associated with catheter-related right internal jugular vein thrombosis in pediatric patients. The study enrolled 80 pediatric patients who were scheduled to receive central venous catheter. To detect thrombus formation, Doppler ultrasound examinations from the thyroid cartilage level to the supraclavicular region were used after CVC placement and on each of the following days until the catheter was removed.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients who were scheduled to catheterize central venous catheter

Exclusion Criteria:

* patients who had skin infections on the right side of the neck, making them unsuitable for placement of the catheter via the right side of the neck
* patients who had blood coagulation lesions or bleeding tendencies
* patients with thrombocytopenia
* patients with a history of right internal jugular vein thrombosis
* patients who presented right internal jugular vein thrombosis or stenosis on preoperative Doppler ultrasound examination

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
thrombus formation using doppler ultrasound examination of internal jugular vein | after central venous catheter placement and on each of the following days until the catheter was removed (maximum 5 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided